CLINICAL TRIAL: NCT05865457
Title: Efficacy and Safety of BUFY02 Versus TRB02 in the Treatment of Dry Eye Disease: a Non-inferiority Investigation
Brief Title: Efficacy and Safety of BUFY02 Versus TRB02 in the Treatment of Dry Eye Disease
Acronym: BUSTON-02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUFY02-CT-2201
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUFY02 (Experimental): 0.3% Sodium Hyaluronate (trometamol buffer) in single-dose containers of 0.45 mL
  Interventions: Device: BUFY02 eye drops in single-dose containers
- TRB02 (Active Comparator): 0.3% Sodium Hyaluronate (phosphate buffer) in single-dose containers of 0.45 mL
  Interventions: Device: TRB02 eye drops in single-dose containers

INTERVENTIONS:
Device: BUFY02 eye drops in single-dose containers — 1 to 2 drops in each eye, as often as needed
  Arms: BUFY02
Device: TRB02 eye drops in single-dose containers — 1 to 2 drops in each eye, as often as needed
  Arms: TRB02

SUMMARY:
The goal of this interventional investigation is to compare BUFY02 with TRB02 in the treatment of patients with dry eye disease. The main questions it aims to answer are:

* Is BUFY02 non-inferior to TRB02 in terms of signs of DED?
* Is BUFY02 non-inferior to TRB02 in terms of symptoms of DED?

Participants will be asked to:

* Visit the trial site at 4 different timepoints
* Use the allocated study treatment everyday until the end of the study (during 3 months)
* Be examined by the investigator
* Complete several questionnaires
* Return unused study treatment.

Researchers will compare BUFY02 to TRB02 to see if both study treatments provide similar effects on signs and symptoms of the disease, together with comparable safety.

ELIGIBILITY:
Inclusion Criteria include:

* At least a 3-month documented history of bilateral dry eye syndrome needing artificial tears;
* At least one eye with Oxford score ≥ 4 and ≤ 9;
* At least one objective sign of tear deficiency (in at least one eligible eye);
* Having a health insurance.

Exclusion Criteria include:

* Wear of contact lenses starting within the last 2 months;
* Best-corrected visual acuity (BCVA) < 1/10;
* Severe DED with one of the listed conditions:
* Severe blepharitis;
* Seasonal allergy;
* Any issues of the ocular surface not related to DED;
* History of ocular trauma, infection or inflammation not related to DED;
* History of ocular surgery, including laser surgery;
* Unstable glaucoma;
* Use of artificial tears with preservative within the last 2 weeks;
* Systemic (enteral or parenteral) or local (topical) use of one of the listed medications:
* Known hypersensitivity to any constituent of the study treatments;
* Pregnancy or breastfeeding;
* Participation in another clinical study within the last 90 days;
* Legally restricted autonomy, freedom of decision and action.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Signs | Day 28
  Change from baseline in Oxford score (0-15, a higher score meaning a worse outcome)

SECONDARY OUTCOMES:
Symptoms | Day 28
  Change from baseline in Ocular Surface Disease Index

CONTACTS AND LOCATIONS:
Locations (5):
- Austria (2):
  - Medical University Graz, Graz
  - VIROS, Vienna
- France (3):
  - CHRU Brest, Brest
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Nice, Nice

IPD SHARING:
Plan to Share IPD: No